CLINICAL TRIAL: NCT04877457
Title: A Phase 4, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Assess the Efficacy of Ocrelizumab in Patients With Radiologically Isolated Syndrome
Brief Title: Ocrelizumab for Preventing Clinical Multiple Sclerosis in Individuals With Radiologically Isolated Disease.
Acronym: CELLO
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: Yale University (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Erin E Longbrake, Assistant Professor of Neurology, Yale University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2000029952; ML42790 (Other: Genentech, Inc.)
Record Dates: First submitted 2021-04-30; First posted 2021-05-07 (Actual); Results first posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Radiologically Isolated Syndrome; Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — ocrelizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomization and blinding will be employed to minimize bias in treatment assignment and to provide the basis for valid statistical inference.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ocrelizumab (Experimental): Three courses of ocrelizumab will be administered over the course of the study.
  Interventions: Drug: Ocrelizumab
- Placebo (Placebo Comparator): Three courses of placebo will be administered over the course of the study.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Ocrelizumab — The first course of ocrelizumab will be administered as two 300 mg infusions at Week 0 (Day 1) and Week 2 (Day 15), with the subsequent second- and third-courses given as a single 600 mg infusion at Weeks 24 and 48.
  Arms: Ocrelizumab
Other: Placebo — Placebo will be administered at Week 0 (Day 1) and Week 2 (Day 15), with the subsequent second- and third-courses given at Weeks 24 and 48.
  Arms: Placebo

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled, Phase 4 study in which eligible patients with RADIOLOGICALLY ISOLATED SYNDROME (RIS) (as defined by meeting 2017 McDonald criteria for DIS) will be randomized 1:1 to receive ocrelizumab treatment or placebo (standard of care).

DETAILED DESCRIPTION:
This study is designed to investigate the treatment effect of ocrelizumab compared with placebo on clinical and radiological outcomes in patients with RIS (i.e., asymptomatic CNS lesions fulfilling the 2017 McDonald criteria for DIS), as well as neuroimaging, serologic, immunologic and other exploratory biomarkers of MS disease biology in order to improve the understanding of B cell biology in early disease pathophysiology, characterize the emergence of CNS autoimmunity, and the mechanism of action of ocrelizumab in this population.

ELIGIBILITY:
Inclusion Criteria

Pre-Screening of First-Degree Family Members

Family members must meet the following inclusion criteria for pre-screening:

Signed informed consent form First-degree family member of an individual with clinically definite MS Age 18-55 years No prior exposure to DMT or long-term immunomodulatory medications Willingness to participate in full study protocol, if RIS is discovered

Screening

Patients must meet the following inclusion criteria for screening:

Signed informed consent form

One of the following:

First degree family member of an individual with clinically definite MS who was identified to have CNS lesions meeting McDonald 2017 criteria for DIS during a pre-screening MRI.

Established RIS diagnosis (i.e. CNS lesions consistent with MS, meeting McDonald 2017 criteria for DIS), either diagnosed within the last 5 years or known to have had accumulation of CNS lesions within the last 5 years.

Age 18-55 years No prior exposure to DMT or long-term immunomodulatory medications Willingness to participate in full study protocol

Randomization

Patients must meet the following criteria for study entry and randomization:

Signed Informed Consent Form Aged 18-55 years at time of signing Informed Consent Form Ability to provide written informed consent and be compliant with the study protocol CNS lesions consistent with MS, meeting McDonald 2017 criteria for DIS RIS diagnosis established within last 5 years OR with known accumulation of CNS lesions within last 5 years No alternative diagnosis established during serologic workup for MS mimics Women of childbearing potential must agree to remain abstinent (refrain from heterosexual intercourse) or use one method of contraception with a failure rate of <1% per year or a barrier method supplemented with spermicide. Contraception must continue for the duration of study treatment and for at least 24 weeks after the last dose of study treatment.

* A woman is considered to be of childbearing potential if she is postmenarcheal, has not reached a postmenopausal state (≥ 12 continuous months of amenorrhea with no identified cause of other than menopause), and has not undergone surgical sterilization (removal of the ovaries and/or uterus)
* Examples of contraceptive methods with a failure rate of <1% per year include bilateral tubal ligation, male sterilization, established hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices.
* The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence and withdrawal are not acceptable methods of contraception.
* Examples of barrier methods supplemented with the use of spermicide include male or female condom, cap, diaphragm, or sponge.

Exclusion Criteria

Patients who meet any of the following criteria will be excluded from pre-screening, screening and randomization:

Intolerance to gadolinium-based contrast agent Contraindications to MRI 5 years of radiologic stability since first known abnormal MRI, for patients previously diagnosed with RIS History of remitting clinical symptoms consistent with MS lasting 24 hours prior to CNS imaging revealing anomalies suggestive of MS CNS MRI anomalies are better accounted for by another disease process, for patients previously diagnosed with RIS Infection Related Known presence of recurrent or chronic infection (e.g., HIV, syphilis, tuberculosis) History of recurrent aspiration pneumonia requiring antibiotic therapy History or known presence of infectious causes of myelopathy (e.g., syphilis, Lyme disease, HTLV-1, herpes zoster myelopathy) Known active bacterial, viral, fungal, mycobacterial infection, or other infection (including tuberculosis or atypical mycobacterial disease, but excluding fungal infection of nail beds) or any major episode of infection requiring hospitalization or treatment with IV antibiotics within 4 weeks prior to baseline visit or oral antibiotics within 2 weeks prior to baseline visit Cancer Related History of cancer, including solid tumors and hematological malignancies (except basal cell, in situ squamous cell carcinomas of the skin, and in situ carcinoma of the cervix or the uterus that have been excised and resolved with documented clean margins on pathology) Pregnant or lactating, or intending to become pregnant during the treatment phase and 6 months after the last infusion of study drug Women of childbearing potential must have a negative serum or urine pregnancy test result within 14 days prior to initiation of study drug.

Other Medical Conditions History of or currently active primary or secondary immunodeficiency History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies History of alcohol or other drug abuse within 24 weeks prior to enrollment History or known presence of systemic autoimmune disorders associated with systemic symptoms (e.g., lupus, anti-phospholipid antibody syndrome, Sjögren's syndrome, Behçet's disease) Any concomitant disease that may require chronic treatment with systemic corticosteroids or immunosuppressants during the course of the study Significant, uncontrolled disease, as defined by AMA guidelines or similar, such as cardiovascular (including congestive heart failure - NYHA grade 3 or 4, cardiac arrhythmia), uncontrolled hypertension, pulmonary (including chronic obstructive pulmonary disease), renal, hepatic, endocrine (including uncontrolled diabetes mellitus), gastrointestinal, or any other significant disease

Known presence or history of other neurologic disorders, including but not limited to, the following:

Progressive multifocal leukoencephalopathy, CNS or spinal cord tumor, potential metabolic causes of myelopathy (e.g., untreated vitamin B12 deficiency) History of genetically inherited progressive CNS degenerative disorder (e.g., hereditary paraparesis; mitochondrial encephalopathy, lactic acidosis, and stroke-like episodes [MELAS]) Neuromyelitis optica spectrum disorders (NMOSD) Ischemic cerebrovascular disorders (e.g., stroke, transient ischemic attack) or ischemia of the spinal cord Severe, clinically significant brain or spinal cord trauma (e.g., cerebral contusion, spinal cord compression) Psychosis not yet controlled by a treatment Drug Related Systemic, high dose corticosteroid therapy within 4 weeks prior to screening Contraindications for, or intolerance to, oral or IV corticosteroids, including IV methylprednisolone, according to the country label, including hypersensitivity to any of the treatment drug constituents Prior exposure to immunomodulatory medications and/or DMT Prior treatment with any disease modifying therapy for MS including but not limited to: interferon (IFN-β-1a (Avonex, Rebif), IFN-β-1b (Betaseron/Betaferon), glatiramer acetate, dimethyl fumarate (DMF; Tecfidera), diroximel fumarate (Vumerity) fingolimod (Gilenya) or siponimod (Mayzent), ozanimod (Zeposia®) natalizumab (Tysabri), alemtuzimab (Lemtrada), cladribine (Mavenclad), rituximab (Rituxan), and other anti-CD20 agents Previous treatment with cyclophosphamide, mitoxantrone, azathioprine, mycophenolate mofetil, cyclosporine, methotrexate, total body irradiation, or bone marrow transplantation Previous or concurrent treatment with any investigational agent or treatment with any experimental procedure for MS (e.g., treatment for chronic cerebrospinal venous insufficiency) Vaccinations: Receipt of a live or live-attenuated vaccine or an inactivated/non-live vaccine within 6 weeks prior to enrollment

Laboratory: Certain laboratory abnormalities or findings at screening, including the following:

Positive serum β-hCG Positive for hepatitis B (hepatitis B surface antigen [HBsAg] positive or hepatitis B core antibody [total HBcAb] confirmed by positive viral DNA polymerase chain reaction [PCR]) AST or ALT less than or equal to 3.0, upper limit of normal Total white blood cell count, including differential counts, below lower limit of normal Absolute lymphocyte count below lower level of normal Absolute neutrophil count below lower limit of normal Platelet count below lower limit of normal

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2023-06-12 (Actual); Study Completion 2023-06-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Yale University, North Haven, Connecticut
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Cleveland Clinic Melen Center, Cleveland, Ohio
  - Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Longbrake EE, Hua LH, Mowry EM, Gauthier SA, Alvarez E, Cross AH, Pei J, Priest J, Raposo C, Hafler DA, Winger RC. The CELLO trial: Protocol of a planned phase 4 study to assess the efficacy of Ocrelizumab in patients with radiologically isolated syndrome. Mult Scler Relat Disord. 2022 Dec;68:104143. doi: 10.1016/j.msard.2022.104143. Epub 2022 Aug 22. PMID 36031693

RESULTS

PARTICIPANT FLOW:
Groups:
- Ocrelizumab - Participants Without a First Degree Family Member With Multiple Sclerosis: Three courses of ocrelizumab will be administered over the course of the study.
  Ocrelizumab: The first course of ocrelizumab will be administered as two 300 mg infusions at Week 0 (Day 1) and Week 2 (Day 15), with the subsequent second- and third-courses given as a single 600 mg infusion at Weeks 24 and 48.
- Placebo - Participants Without a First Degree Family Member With Multiple Sclerosis.: Three courses of placebo will be administered over the course of the study.
  Placebo: Placebo will be administered at Week 0 (Day 1) and Week 2 (Day 15), with the subsequent second- and third-courses given at Weeks 24 and 48.
Period: Overall Study
Arm/Group | Ocrelizumab - Participants Without a First Degree Family Member With Multiple Sclerosis | Placebo - Participants Without a First Degree Family Member With Multiple Sclerosis.
Started | 2 | 1
Completed | 0 | 0
Not Completed | 2 | 1
Not completed — Early termination of study due to low enrollment | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ocrelizumab | Placebo | Total
Number analyzed (Participants) | 2 | 1 | 3
Age, Continuous [Mean (Full Range); unit: Years] | 31 [27 to 35] | 35 [35 to 35] | 33 [27 to 35]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 1 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Smoking status [Count of Participants; unit: Participants] | 0 | 0 | 0
History of infectious mononucleosis [Count of Participants; unit: Participants] | 1 | 0 | 1
History of childhood/adolescent obesity [Count of Participants; unit: Participants] | 1 | 0 | 1
Number of participants with a family history of MS [Count of Participants; unit: Participants] | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Time to Development of First New Radiologic or Clinical Evidence of MS
Description: The primary efficacy endpoint for this study is to evaluate the efficacy of ocrelizumab compared with placebo on delaying the time to development of new radiological or clinical evidence of MS, defined as the time from baseline to first new T1 gadolinium-enhancing lesions and/or new or enlarging T2 lesions consistent with MS in participants OR first clinical evidence of MS, i.e., neurological event resulting from CNS demyelination as evidenced by acute or progressive clinical syndrome consistent with MS in participants.
Time Frame: Up 4 years
Population: Data not collected due to early termination of study
Arm/Group | Ocrelizumab | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Cumulative Number of New or Enlarging T2 Lesions
Description: MRI scans will be used to determine the number of new or enlarging T2 lesions
Time Frame: Up to 4 years
Population: Data for this outcome was not collected.
Arm/Group | Ocrelizumab | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Change in T2-lesion Volume
Description: MRI scans will be used to the change in T2 lesions
Time Frame: Baseline, 24 weeks, 48 weeks, 72 weeks, 104 weeks, 156 weeks, 208 weeks
Population: Data for this outcome was not collected.
Arm/Group | Ocrelizumab | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Cumulative Number of New T1 Gadolinium-enhancing Lesions
Description: MRI scans will be used to determine the cumulative number of new T1 gadolinium-enhancing lesions
Time Frame: Up to 4 years
Population: Data for this outcome was not collected.
Arm/Group | Ocrelizumab | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change in Total Brain Volume
Description: MRI scan will be used to determine the change in total brain volume
Time Frame: Baseline, 24 weeks, 48 weeks, 72 weeks, 104 weeks, 156 weeks, 208 weeks
Population: Data for this outcome was not collected.
Arm/Group | Ocrelizumab | Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Change in Total Spinal Cord Volume
Description: MRI scan will be used to determine the change in total brain volume
Time Frame: Baseline, 24 weeks, 48 weeks, 72 weeks, 104 weeks, 156 weeks, 208 weeks
Population: Data for this outcome was not collected.
Arm/Group | Ocrelizumab | Placebo
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Change in Serum NfL (sNfL)
Description: Change in serum Nfl will be used measured
Time Frame: Baseline, 24 weeks, 48 weeks, 72 weeks, 104 weeks, 130 weeks, 156 weeks, 182 weeks, 208 weeks
Population: Data for this outcome was not collected.
Arm/Group | Ocrelizumab | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: The period of time over which adverse event data were collected was over one year.
Description: All adverse events were not study-drug related. The total number of subjects therefore not at risk for the adverse events that occurred and were reported.
Arm/Group | Ocrelizumab | Placebo
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/1
Other Adverse Events (participants affected / at risk) | 1/2 | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ocrelizumab (N=2) | Placebo (N=1)
Positional headache (General disorders) | 0 | 1 (1) — Positional headache following lumbar puncture. Headache lasted for three days and was treated with an epidural blood patch. Issue was resolved.
Blurry vision (Eye disorders) | 0 | 1 (1) — Subject experienced blurry vision and was referred to neuroophthalmologist and MRI of the orbits was ordered. Subject was diagnosed with astigmatism. Issue is ongoing.
Left ear infection (Ear and labyrinth disorders) | 1 (1) | 0 (0) — Subject experienced a left ear infection. Treated with fluticasone E prop 50mcg spray BID, Amoxicillin Clavulanate 1 tab BID, Claritin D 24 hr 10mg QD. Issue resolved and not related to study drug.

LIMITATIONS AND CAVEATS:
Early termination leading to small number of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-22): https://cdn.clinicaltrials.gov/large-docs/57/NCT04877457/Prot_SAP_000.pdf